CLINICAL TRIAL: NCT01592929
Title: Assessment of the Effect of the Shape of an Inhaler's Mouthpiece on Upper Airway Geometry, Using Functional Respiratory Imaging and Pharyngometry.
Brief Title: Evaluation With Scans and Pharyngometry of the Possible Changes in Upper Airway Geometry Induced by Using Different Mouthpieces.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FLUIDDA nv (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FLUI-2011-80
Record Dates: First submitted 2012-05-04; First posted 2012-05-07 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2012-11

CONDITIONS: Influence of Mouthpiece Design on Upper Airway Geometry
Keywords: Functional Respiratory Imaging; Magnetic Resonance Imaging; MRI; Pharyngometry; Upper Airway; Mouthpiece of Inhaler; Cone Beam Computed Tomography; CBCT; Computed Tomography; CT
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Dental Impression Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Magnetic Resonance imaging — 11 MRI scans per subject will be taken, one for each mouthpiece design of an inhaler.
  Other Names: MRI
Other: Pharyngometry — Pharyngometry will be carried out in supine and upright position. 11 different mouthpieces will be evaluated in both positions.
Radiation: Computed Tomography scan — One low dose CT scan of the upper airway will be taken. The scan will be taken at normal inhalation through a mouthpiece with moderate resistance.
  Other Names: CT scan
Radiation: Cone Beam Computed Tomography scan — One CBCT scan of the upper airway will be taken. The scan will be taken at normal respiration through a mouthpiece with moderate resistance.
  Other Names: CBCT scan
Other: Dental impressions — Dental impressions will be taken. These will be optically scanned before registration in the 3D imaging modalities.

SUMMARY:
In this study the possible changes in upper airway geometry induced by variations in the characteristics of the mouthpieces of inhalers will be evaluated with functional respiratory imaging (FRI) and Pharyngometry. The study population consists of 12 healthy male subjects.

Different mouthpiece designs will be evaluated for each subject by using magnetic resonance imaging (MRI) scans. The results will help to identify the influence of the height, width, protrusion and resistance of the mouthpiece on upper airway geometry.

Pharyngometry profiles of all subjects, whilst inhaling through different mouthpiece variants, in supine and upright position, will be completed.

A computed tomography (CT) scan and a cone beam computed tomography (CBCT) scan of the upper airway will be taken to respectively compare the time dependence on 3D imaging with MRI and to provide a 3D image in an upright position.

Dental impressions will be optically scanned to obtain a more accurate representation of the oral cavity, mainly in MRI.

ELIGIBILITY:
Inclusion Criteria:

* Male subject ≥ 18 years old
* Written informed consent obtained
* BMI ≥ 20 kg/m2 and < 25 kg/m2
* Height ≥ 175 cm and ≤ 185 cm
* Subject must be able to understand and complete the protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

* Subject with claustrophobia
* Subject with a history of surgery of the upper airway
* Subject with an enlarged thyroid gland
* Subject with intra-oral piercings
* Subject with dental bracket
* Subject with a pacemaker or another implant that is likely to interfere with the MRI procedure
* Subject that is unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study
* Subject who received any investigational new drug within the last 4 weeks prior to visit 1.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Changes in upper airway geometry by using MRI. | Within 20 days after day 1
  The primary objective of this study is to evaluate with MRI-FRI the possible changes in upper airway geometry induced by using different mouthpieces.

SECONDARY OUTCOMES:
Changes in upper airway geometry by using pharyngometry in supine versus upright position. | Within 20 days after day 1
  Secondary the assessment of the effect of using different mouthpieces on changes in upper airway geometry by using pharyngometry in supine versus upright position will be performed.

OTHER OUTCOMES:
Evaluate time dependence on image upper airway by using CT scan | At day 1
  With a high resolution computed tomography (HRCT) scan it's possible to obtain high resolution images in a very short period of time at a low radiation dose. Therefore the 3D CT image of the upper airway will be compared with the one from MRI for 1 mouthpiece to check the time dependence. MRI takes about 50 seconds and CT only 3-4 seconds.
3D image of upper airway in upright position by using CBCT scan | At day 1
  To make a comparison between the upright and supine upper airway geometry the CBCT will be used to provide a 3D image of the upper airway in an upright position. This image will be compared with the 3D MRI image for 1 mouthpiece.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Backer, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium